CLINICAL TRIAL: NCT02471521
Title: Optimal Inspiratory Pressure for Facemask Pressure-controlled Ventilation in Children: Study Using Detection of Gastric Insufflation Using Ultrasonography of the Antrum and Epigastric Auscultation
Brief Title: Optimal Inspiratory Pressure for Facemask Pressure-controlled Ventilation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, associated professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1412-083-633
Record Dates: First submitted 2015-06-06; First posted 2015-06-15 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Child; Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuromuscular blocker (Experimental): During induction of anesthesia, mask ventilation by pressure controlled ventilation is performed with after rocuronium administration in children while continuous gastric auscultation and abdominal sonography are performed.
  Interventions: Other: Mask ventilation; Drug: Rocuronium
- Non-neuromuscular blocker (Active Comparator): During induction of anesthesia, mask ventilation by pressure controlled ventilation is performed without rocuronium in children while continuous gastric auscultation and abdominal sonography are performed.
  Interventions: Other: Mask ventilation

INTERVENTIONS:
Other: Mask ventilation — Mask ventilation is performed after administration of rocuronium or not. Initial inspiratory pressure is set as 10 cmH2O and increased gradually by 2 cmH2O until gastric insufflation is detected by either of two methods. Tracheal intubation is done after detection of gas.
Drug: Rocuronium — Rocuronium 0.6 mg/kg is injected before mask ventilation in muscle relaxant group or after finish of study in non-relaxant group.
  Arms: Neuromuscular blocker

SUMMARY:
The purpose of this study is to find an optimal inspiratory pressure to provide adequate tidal volume and prevent gastric insufflation in pediatric patients.

The children under 5 years old are randomly assigned to muscle relaxation group and non-relaxation group. For muscle relaxation group, routine anesthesia induction is performed with muscle relaxant and mask ventilation is started by pressure-controlled mechanical ventilation. Gastric auscultation and abdominal ultrasonography are performed simultaneously during mask ventilation to detect inflow of air. Initial inspiratory airway pressure is 10 cmH2O and increased gradually by 2 cmH2O until gastric insufflation is detected by either of two methods. Tracheal intubation is done after detection of gas.

For non-relaxation group, mask ventilation is performed in a same manner, without muscle relaxant. After detection of gas by any of the two methods, rocuronium 0.6 mg/kg is administered and tracheal intubation is performed.

DETAILED DESCRIPTION:
The purpose of this study is to find an optimal inspiratory pressure to provide adequate tidal volume and prevent gastric insufflation in pediatric patients.

The children under 5 years old are randomly assigned to muscle relaxation group and non-relaxation group. Stratum was constructed based on age and randomization scheme was performed separately within each stratum. Block randomization was done to ensure balance of the age groups.

For muscle relaxation group, routine anesthesia induction is performed with muscle relaxant and mask ventilation is started by pressure-controlled mechanical ventilation. Gastric auscultation and abdominal ultrasonography are performed simultaneously during mask ventilation to detect inflow of air. Initial inspiratory airway pressure is 10 cmH2O and increased gradually by 2 cmH2O until gastric insufflation is detected by either of two methods. Tracheal intubation is done after detection of gas.

For non-relaxation group, mask ventilation is performed in a same manner, without muscle relaxant. After detection of gas by any of the two methods, rocuronium 0.6 mg/kg is administered and tracheal intubation is performed.

Tidal volume and oxygen saturation are recorded during study period.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for elective surgery under general anesthesia
* BMI < 30
* ASA class 1 or 2

Exclusion Criteria:

* with difficult airway
* preexisting pulmonary disease
* upper respiratory tract infection
* intestinal obstruction
* with risk of pulmonary aspiration
* history of stoke or moyamoya disease

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD. PhD., Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JH, Jung H, Kim EH, Song IK, Kim HS, Kim JT. Optimal inspiratory pressure for face mask ventilation in paralyzed and unparalyzed children to prevent gastric insufflation: a prospective, randomized, non-blinded study. Can J Anaesth. 2018 Dec;65(12):1288-1295. doi: 10.1007/s12630-018-1183-2. Epub 2018 Jul 11. PMID 29998359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center study was performed in a tertiary children's hospital in Republic of Korea.
Groups:
- Neuromuscular Blocker Group: Facemask ventilation was performed after rocuronium (0.6mg/kg) was administered.
- Non-neuromuscular Blocker Group: Facemask ventilation was performed without rocuronium administration.
Period: Overall Study
Arm/Group | Neuromuscular Blocker Group | Non-neuromuscular Blocker Group
Started | 60 | 60
Completed | 60 | 52
Not Completed | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Blocker Group | Non-neuromuscular Blocker Group | Total
Number analyzed (Participants) | 60 | 52 | 112
Age, Continuous [Mean (Full Range); unit: years] | 1.2 [0.1 to 5.0] | 1.4 [0.1 to 4.0] | 1.3 [0.1 to 5.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 39 | 31 | 70
Height [Mean (Standard Deviation); unit: cm] | 76.0 (14.3) | 78.8 (14.2) | 77.2 (14.5)
Weight [Mean (Standard Deviation); unit: kg] | 10.0 (3.8) | 10.4 (3.5) | 10.3 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Pressure That Cause Gastric Insufflation
Description: Difference in the inspiratory pressure that minimized the incidence of gastric insufflation, yet guaranteed a tidal volume of at least 6 ml/kg between the neuromuscular blocker and non-neuromuscular blocker groups.
  Gastric insufflation was measured using both gastric ultrasonography and epigastric auscultation.
Time Frame: Interval between start of mask ventilation and detection of gastric insufflation, an expected average of 100 sec
Measure: Mean (Full Range); unit: cmH2O
Arm/Group | Neuromuscular Blocker Group | Non-neuromuscular Blocker Group
Number analyzed (Participants) | 60 | 52
cmH2O | 13 [12 to 14] | 13 [12 to 14]

2. Secondary Outcome: Diagnostic Method That Detects Gastric Insufflation First
Time Frame: Interval between start of mask ventilation and detection of gastric insufflation, an expected average of 100 sec
Measure: Count of Participants; unit: Participants
Arm/Group | Neuromuscular Blocker Group | Non-neuromuscular Blocker Group
Number analyzed (Participants) | 60 | 52
Participants
  Ultrasound | 44 | 23
  Auscultation | 4 | 10
  Simultaneous detection by both methods | 12 | 19

ADVERSE EVENTS:
Arm/Group | Neuromuscular Blocker Group | Non-neuromuscular Blocker Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/52
Other Adverse Events (participants affected / at risk) | 0/60 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No